CLINICAL TRIAL: NCT01569061
Title: A Double-blind, Randomized, Sham-controlled, Multicenter Clinical Trial to Assess the Effectiveness of Therapeutic Class IV Laser LCT-1000TM Treatment for Overactive Bladder Syndrome.
Brief Title: Painless Laser Therapy for Overactive Bladder
Acronym: PLTOAB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zipper Urogynecology Associates (Other)
Responsible Party: Principal Investigator, Ralph Zipper, MD, Principal Investigator, Zipper Urogynecology Associates
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11-179
Record Dates: First submitted 2012-03-26; First posted 2012-04-02 (Estimated); Last update posted 2012-04-02 (Estimated); Status verified 2012-03

CONDITIONS: Overactive Bladder
Keywords: overactive bladder; laser therapy; urinary incontinence; urinary urgency
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Laser Group (ALG) (Active Comparator)
  Interventions: Device: LCT-1000TM (Manufacturer: LiteCure)
- Sham Laser Group (SLG) (Sham Comparator)
  Interventions: Device: LCT-1000TM (Manufacturer: LiteCure)

INTERVENTIONS:
Device: LCT-1000TM (Manufacturer: LiteCure) — low level laser therapy (LLLT)
  Arms: Active Laser Group (ALG)
Device: LCT-1000TM (Manufacturer: LiteCure) — low level laser therapy (LLLT) sham treatment
  Arms: Sham Laser Group (SLG)

SUMMARY:
The primary objective of this study is to determine the effectiveness of transvaginally-delivered low level laser therapy (LLLT) versus Sham in the treatment of overactive bladder symptoms in women. The secondary objective is to determine the effect of transvaginally-delivered LLLT vs. sham on the quality of life.

DETAILED DESCRIPTION:
This study is a double-blind, randomized, sham-controlled, multicenter, clinical trial that will include enrollment of up to 200 subjects at up to 3 investigational sites.

The study population will be randomized at a 1:1 ratio into two groups: Sham Laser Group (SLG) and Active Laser Group (ALG). The Sham Laser Group will receive a sham LLLT procedure (no laser energy) and the Active Laser Group will receive an active LLLT procedure (laser energy).

Both groups will undergo 3 LLLT procedures per week for 3 weeks, for a total of 9 LLLT procedures. Whether the procedure will be a sham procedure (placebo) or an active LLLT application will be determined by randomization which will assign subjects to be treated with an LCT-1000TM labeled either Laser A or Laser B. The only difference between Laser A and Laser B is that one does not emit laser energy; therefore, both subjects and site research personnel will be blinded as to whether laser energy is actually applied to the subject.

ELIGIBILITY:
Inclusion Criteria:

* The subject is female and at least 18 years of age at screening.
* A score of > 4 on the OAB-q short form for urgency.
* The subject has an average urinary frequency of > 10 voids per day.
* Self-reported bladder symptoms for > 3 months.
* Self-reported failed conservative care.
* The subject has discontinued all antimuscarinics for at least 2 weeks prior to screening.
* The subject is ambulatory and able to use the toilet independently and without difficulty.
* Negative pregnancy test in subjects of childbearing potential.
* Subject attests in writing that she has not had unprotected intercourse within 3 weeks prior to study enrollment and agrees to have no intercourse until treatments conclude.
* Subject Informed Consent obtained in writing in compliance with local regulations prior to enrollment into this study.
* The subject (and caregiver, if applicable) is willing to participate in this study for at least 7 weeks.
* The subject is otherwise in general good health with no other major medical conditions.

Exclusion Criteria:

* The subject has vaginal bleeding.
* The subject has urinary or gastric retention or a neurogenic bladder.
* The subject is not capable of completing study questionnaires or undergoing portions of the study.
* The subject has been sexually assaulted.
* The subject has an alcohol or drug addiction.
* The subject has used isotretinoin (Accutane) within 6 months prior to study enrollment.
* The subject has cancer.
* The subject has used Botox® in the bladder or pelvic floor muscles within 12 months prior to study enrollment.
* The subject currently has a urinary tract infection or vaginal infection.
* The subject is using Interstim® or Bion®.
* Current use of TENS in pelvic region, back or legs.
* The subject is pregnant or lactating, or is of childbearing potential unless she is surgically sterile or she and/or her partner are using a medically acceptable method of birth control.
* Any use of light-activated drugs (photodynamic therapy) or heat sensitive medications within 30 days of first treatment.
* The subject has used an investigational drug/device therapy or participated in any clinical investigation involving or impacting gynecologic, urinary, or renal function within 4 weeks prior to study enrollment.
* The subject is otherwise determined, based on the opinion of the Investigator, to be an unsuitable candidate for enrollment in this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-02; Primary Completion 2013-08 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy endpoint will be the improvement of OAB symptoms and general quality of life due to the effect of LLLT treatment on OAB through week 7. | Visits 3, 4, 5, 6, 7, 8, 9, 10, 11, 12 and 13 (over approximately 7 weeks)
  Patients will undergo 3 LLLT procedures per week for 3 weeks, for a total of 9 LLLT procedures.
The primary safety endpoint will evaluate the SLG and ALG treatment groups for differences in reported side effects and adeverse events throughout the trial, including LLLT treatment and follow-up. | Visits 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12 and 13 (over approximately 8 weeks)
  Patients will undergo 3 LLLT procedures per week for 3 weeks, for a total of 9 LLLT procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Zipper, MD, Principal Investigator — Zipper Urogynecology Associates
Locations (1):
- Zipper Urogynecology Associates, Melbourne, Florida, United States

REFERENCES:
- See also: Zipper Urogynecology Associates — http://www.zipperurogyn.com/